CLINICAL TRIAL: NCT03148184
Title: Reverse Shoulder Arthroplasty in Patients 60 Years Old and Younger: Short-term Clinical and Radiographic Results
Brief Title: Reverse Shoulder Replacement: Age 60 or Younger Outcomes
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 201408124
Record Dates: First submitted 2017-03-08; First posted 2017-05-10 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Shoulder Arthritis
Keywords: reverse total shoulder arthroplasty; 60 years old or younger; outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: shoulder x-ray — post operative shoulder x-ray at minimum 2 year post op

SUMMARY:
The purpose of this study is to assess the early outcomes following Reverse Shoulder Arthroplasty (RSA) in patients sixty years or younger for the purpose of characterizing these patients, evaluating their clinical outcomes and radiographic appearance.The investigators would like to know how quickly they are healing and returning to their baseline activities of daily living and ability to work. This will help when counseling patients prior to surgery as it will give us a better defined and study supported understanding of the post-operative recovery timeline in the younger population.

DETAILED DESCRIPTION:
This study is looking at patients who are sixty years or younger at the time of they undergo a reverse total shoulder replacement. This is an important population to look at their functional and clinical outcomes as they are often still employed and have more physical demands upon their shoulder in everyday life than the older replacement population for which there are more outcome data available. The investigators would like to determine how the younger population is healing and returning to their baseline activities of daily living and ability to work. This will help when counseling patients prior to surgery as it will give us a study supported understanding of the post-operative recovery timeline in the younger population. The investigators will review x-rays to evaluate healing at two years. Functional surveys are given pre and post operatively (1 & 2 years) and these will be reviewed as well. A physical exam is also performed to determine range of motion pre and post operatively (1 & 2 years).

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or younger at the time of surgery
* reverse shoulder arthroplasty with a single implant system by one of our four surgeons

Exclusion Criteria:

* minors
* unable to complete imaging portion of the two-year follow-up due to health safety/exposure concerns
* unwilling/unable to return for follow up
* Revision procedure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients age 60 or younger who are will undergo or have undergone a primary reverse shoulder arthroplasty with a single implant system by one of our four surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Assess functional change from before surgery to two years post surgery | 2 years post op
  Assess changes in range of motion as part of the overall clinical outcome function scores. ASES (American Shoulder and Elbow Questionnaire)

SECONDARY OUTCOMES:
Radiographic Outcomes | 2 years post op
  Evaluate the shoulder replacement for any signs of implant loosening or bone loss. X-rays are reviewed by Orthopedic Surgeons. There is either loosening present/absent and bone loss present/absent.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Chamberlain, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frankle M, Levy JC, Pupello D, Siegal S, Saleem A, Mighell M, Vasey M. The reverse shoulder prosthesis for glenohumeral arthritis associated with severe rotator cuff deficiency. a minimum two-year follow-up study of sixty patients surgical technique. J Bone Joint Surg Am. 2006 Sep;88 Suppl 1 Pt 2:178-90. doi: 10.2106/JBJS.F.00123. PMID 16951091
- [Background] Naveed MA, Kitson J, Bunker TD. The Delta III reverse shoulder replacement for cuff tear arthropathy: a single-centre study of 50 consecutive procedures. J Bone Joint Surg Br. 2011 Jan;93(1):57-61. doi: 10.1302/0301-620X.93B1.24218. PMID 21196544
- [Background] Nolan BM, Ankerson E, Wiater JM. Reverse total shoulder arthroplasty improves function in cuff tear arthropathy. Clin Orthop Relat Res. 2011 Sep;469(9):2476-82. doi: 10.1007/s11999-010-1683-z. PMID 21116759